CLINICAL TRIAL: NCT05154838
Title: Development of Volatile Organic Compounds (VOC) Analysis as a Potential Diagnostic for Infected and Non-Healing Wounds
Acronym: AROMA
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Cardiff Metropolitan University (Other)
Responsible Party: Sponsor
Other Study IDs: 7864; 302788 (Other: IRAS)
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2022-03

CONDITIONS: Pilonidal Abscess; Non-healing Wound
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Pilonidal Abcess: All adult (18+) patients presenting at surgical assessment unit requiring treatment for pilonidal abscess. Wounds will be drained, cleaned and packed as per usual clinical practice. Extra standard wound swabs will be collected for additional microbiological analyses. Control wound dressings will be placed on adjacent, unaffected area of skin for 24 hours.
  Interventions: Procedure: Drainage and packing of pilonidal abscess

INTERVENTIONS:
Procedure: Drainage and packing of pilonidal abscess — Patients will be treated as per standard care, their wound drained, cleaned and packed. Microbiology swab samples will be obtained.

SUMMARY:
The study aims to assess the feasibility of detecting volatile organic compounds (VOCs) from pilonidal wound dressings to assemble a VOC profile for the assessment of wound healing trends.

Non-healing wounds (NHWs) pose a significant burden to healthcare providers and to affected patients. Difficulties arise in the identification of wounds which are not on a healing trajectory. Early identification allows for proactive management to try and reduce healing time. Recent studies indicate that wound VOCs may have the potential to differentiate between healing and non-healing wounds. This study will use pilonidal abscesses for the analysis of wound VOC profiles using a non-invasive technique.

DETAILED DESCRIPTION:
Non-healing wounds (NHWs) are a worldwide and costly problem. Although NHWs are relatively small in number, the cost associated for care and product use is disproportionately high. A recent study from the United Kingdom suggests that wound care accounts for an estimated £8.3bn, or approximately 5.5% of total NHS healthcare costs (Guest 2017). NHWs can cause pain, stress, isolation, odour, and decreased mobility for the patients and, if the wound remains after more than 12-24 months, further surgery is required which may be radical and disfiguring.

Emergency presentation of pilonidal abscess requires hospitalisation with incision and drainage of the abscess cavity. Complete healing occurs in 60% of patients (Deans GT 1998) and one in five patients represent with recurrent symptoms following emergency surgery (Jensen 1988). Infection and wound breakdown after elective surgery is also relatively common affecting 10-15% of patients (Spivak H 1996), making it a good candidate to studying non-healing wounds.

Patients over the age of 18 who are admitted to hospital with a pilonidal abscess which requires drainage will be eligible for the study. The patient will undergo the standard procedure to drain an abscess, during which time wound swabs will be collected. Additional swabs will be collected for participants in this study, compared to routine care. The wound will be dressed as standard and the same dressing is applied to an area of un-affected skin on the buttock. The dressings are changed the following day, and are handled in such a way that VOC are released and captured from the dressings. These VOC will be sent for analysis using specialist equipment, which will identify VOC profiles that are unique to each sample. Participants will be followed up 30 days later after treatment to assess the wound-healing status, which will in turn be linked back to the VOC profile in order to determine whether associations can be made between the two. The study aims to recruit 12 patients over a 12 month period.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery for acute pilonidal abscess
* Aged 18 or over and able to give informed consent

Exclusion Criteria:

* Patients who are unwilling or unable to provide informed consent
* Patients who are unable to speak adequate English for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients due to undergo acute surgical treatment for pilonidal sinus disease will be invited to participate in this study. A total of 12 patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Volatile Organic Compound detection | 12 months
  Feasibility of detecting VOC from pilonidal wound dressings as determined by mass-spec

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No